CLINICAL TRIAL: NCT00498329
Title: Brain Connectivity and Sensorimotor Integration During Dual/Single Motor Tasks
Brief Title: Brain Function in Performance of Motor Tasks
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070187; 07-N-0187
Record Dates: First submitted 2007-07-07; First posted 2007-07-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-11-18

CONDITIONS: Brain Connectivity
Keywords: fMRI; Electroencephalogram (EEG); Attention; Sensorimotor Integration; Human Brain; Healthy Volunteer; HV

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will examine how the areas in the brain are connected when they are controlling two finger movements at the same time. It will look at how people use what they see to help guide two different movements. This ability, which is important in everyday life, can be a problem for patients with neurological problems.

Healthy right-handed volunteers 18 years of age and older may be eligible for this study. Candidates are screened with a medical history, physical examination and magnetic resonance imaging (MRI) of the brain. MRI uses a strong magnetic field and radio waves to obtain images of body organs and tissues. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. The subject lies on a table that can slide in and out of the scanner, wearing earplugs to muffle loud noises that occur during the scanning.

Participants undergo functional MRI (fMRI). This is a standard MRI that is done while the subject performs skilled finger tasks in response to instructions they see on a screen. Researchers localize brain areas which show activity changes while the tasks are performed. Before the test session begins, subjects complete a questionnaire and have an opportunity to practice the task.

Subjects control the position of one or two cursors on a screen using one or two fingers. They perform tracking or pointing tasks according to what they see on the screen. During the single-task experiment only one task is presented on the screen. During the dual-task experiment, two tasks are presented on the screen. Subjects perform either the single-task or dual-task experiment, but not both. The fMRI lasts about 90 minutes, with subjects asked to lie still during the scan for up to 9 minutes at a time.

After completing the fMRI, subjects are scheduled for a research electroencephalogram (EEG) and magnetoencephalogram (MEG). The test is done while the subject performs tasks so that researchers can learn about the timing of changes in activity in certain brain regions during performance of the same tasks done for the fMRI.

DETAILED DESCRIPTION:
Objective

Using a block design BOLD-fMRI, we want to investigate the connectivity in brain regions when two motor responses are performed in the same time. The designs will be replicated using EEG and MEG to understand the time course of the activated brain network better. It will allow us to map the brain processes involved in sensorimotor integration and attentional sharing.

Study Population

160 individuals subdivided in:

* 110 adult healthy volunteers
* 25 patients with Parkinson Disease
* 25 patients with Focal Hand Dystonia

Design

Two experiments will be performed using MEG, EEG and fMRI techniques. Both experiments will use visuo-motor control tasks. Two motor responses (given by two fingers of the dominant hand) will be simultaneously performed. Experiment 1 will use single motor tasks; Experiment 2 will use dual motor tasks. In both experiments, the attention demands will vary with the execution mode of the motor outputs (competitive or cooperative). In competitive tasks, the visual stimuli will be used to perform two independent motor outputs. In cooperative tasks, the visual stimuli will be used to perform two coupled motor outputs. The effect of the execution mode on brain connectivity will be isolated comparing competitive and cooperative tasks. The sensory information must be associated to the motor command to perform a given motor task: this process is called sensorimotor integration. With both experiments, we will be able to dissociate the network connectivity linked to:

* sensorimotor integration demands for focused attention in a single task,
* sensorimotor integration demands for divided attention in a dual motor task.

After subjects have been properly trained to perform the tasks, they will undergo fMRI scanning MEG and EEG recording. Subjects will perform the tasks presented pseudo-randomly during six sets of 5-minute sessions. We will record their muscular activity via EMG surface electrodes.

Outcome Measures

The primary outcomes are the task-dependent functional connectivity (for fMRI) between areas and coherence (for MEG and EEG) of cerebral sources relative to performance of the tasks. The force control of two fingers in the same time would elicit blood oxygen level dependent (BOLD) signal and electrical brain activity variations in the network involved in manual dexterity. We are interested in studying the connectivity between the homologous motor areas of the two hemispheres, and between prefrontal cortex and parietal cortex, to understand sensorimotor integration processes during competitive and cooperative dual tasks. As a second measure, we are interested in analyzing coherence between MEG-EMG and EEG-EMG signals.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for Healthy Volunteers

* Subjects age from 18 to older.
* Subjects must be right-hand dominant (Edinburgh Handedness Quotient greater than 60), except if they are part of the control group to match left handed patients.
* Subjects willing to abstain from caffeine or alcohol for 48 hours prior to the fMRI scanning and MEG or EEG recording

Inclusion Criteria for PD Patients

* men and women aged 18 to 75 years with DOPA-responsive PD
* modified Hoehn and Yahr grade of 2 to 4 while OFF
* must be on a medical regimen that includes levodopa.
* total dose of levodopa and dopamine agonists (using dopamine equivalents) has to be equal to or more than 300 milligrams per day
* patients willing to abstain from caffeine or alcohol for 48 hours prior to the fMRI scanning and MEG or EEG recording.

Inclusion Criteria for FHD Patients

* Between 18 and 65 years old
* Diagnosed with focal hand dystonia
* patients willing to abstain from caffeine or alcohol for 48 hours prior to the fMRI scanning and MEG or EEG recording

EXCLUSION CRITERIA:

Exclusion Criteria for Healthy Volunteers

* Subjects with any abnormal findings on the neurological exam,
* Subjects who are pregnant (as determined by positive urine pregnancy test) which prevents them having an MRI
* Subjects with any finding on the MRI safety questionnaire which prevents them from safely undergoing an MRI scan
* Subjects with metallic dental fillings which are likely to cause MRI artifacts
* Subjects with any history of brain tumor, stroke, head trauma or a vascular malformation as obtained by history or from imaging studies
* Subjects with any history of a severe medical condition, such as cardiovascular disease, which would prevent them from lying flat for up to 120 minutes
* Subjects without the capacity to give informed consent
* Subjects with claustrophobia or other restrictions which prevent them from undergoing a scan in a confined space for up to 90 minutes

Exclusion Criteria for PD Patients

* Patients with any abnormal findings on the neurological exam, with the exception of neurological findings consistent with Parkinson disease.
* any active psychiatric disease
* concurrent use of tricyclic antidepressants, neuroleptic agents, or any other licit or illicit drugs other than anti-parkinsonian agents that could lower the seizure threshold except for SSRI
* history of pallidotomy
* presence of implanted electrodes and generator for deep brain stimulation
* the study would cause undue risk or stress for reasons such as excessive fatigue, general frailty, or excessive apprehensiveness.
* dementia as assessed by the Folstein's Mini Mental Test Examination (MMSE < 24/30) or mentally impaired patients having no capacity to provide their own consent (the physician establishing the diagnosis and applying UPDRS will evaluate patient's mental capacity using conventional clinical interview)
* Patients who are pregnant (as determined by positive urine pregnancy test) which prevents them having an MRI
* Patients with any finding on the MRI safety questionnaire which prevents them from safely undergoing an MRI scan
* Patients with metallic dental fillings which are likely to cause MRI artifacts
* Patients with surgically or traumatically implanted foreign bodies such as a pacemaker, implanted medical pump, implanted hearing aids, metal plate in the skull, or metal implant in the skull or eyes (other than dental appliances or fillings) that may pose a physical hazard during MRI.
* Patients with any history of brain tumor, stroke, seizures, head trauma or a vascular malformation as obtained by history or from imaging studies.
* Patients with a history of seizures and/or epilepsy
* Patients with any history of a severe medical condition other than PD, such as cardiovascular disease, which would prevent them from lying flat for up to 120 minutes
* Patients without the capacity to give informed consent
* Patients with claustrophobia or other restrictions which prevent them from undergoing a scan in a confined space for up to 90 minutes

Exclusion Criteria for FHD patients

* Patients with any abnormal findings on the neurological exam, with the exception of neurological findings consistent with Focal Hand dystonia
* Subjects with severe focal hand dystonia at rest.
* Patients with mirror dystonia
* Subjects who have had recent (within 3 months) Botulinum Toxin (Botox) injections
* Patients who are on anti-parkinsonian drugs
* Patients who are pregnant (as determined by positive urine pregnancy test) which prevents them having an MRI
* Patients with any finding on the MRI safety questionnaire which prevents them from safely undergoing an MRI scan
* Patients with metallic dental fillings which are likely to cause MRI artifacts
* Patients with surgically or traumatically implanted foreign bodies such as pacemaker, implanted medical pump, implanted hearing aids, metal plate in the skull, or metal implant in the skull or eyes (other than dental appliances or fillings) that may pose a physical hazard during MRI.
* Patients with any history or brain tumor, stroke, seizures, head trauma or a vascular malformation as obtained by history or from imaging studies
* Patients with a history of seizures and/or epilepsy
* Patients with any history of a severe medical condition, other than PD, such as cardiovascular disease, which will prevent them from lying flat for up to 120 minutes.
* Patients without the capacity to give informed consent
* Patients with claustrophobia or other restrictions which prevent them from undergoing a scan in a confined space for up to 90 minutes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2007-07-03; Study Completion 2011-11-18

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Singer W. Synchronization of cortical activity and its putative role in information processing and learning. Annu Rev Physiol. 1993;55:349-74. doi: 10.1146/annurev.ph.55.030193.002025. No abstract available. PMID 8466179
- [Background] Singer W, Gray CM. Visual feature integration and the temporal correlation hypothesis. Annu Rev Neurosci. 1995;18:555-86. doi: 10.1146/annurev.ne.18.030195.003011. No abstract available. PMID 7605074
- [Background] von der Malsburg C, Schneider W. A neural cocktail-party processor. Biol Cybern. 1986;54(1):29-40. doi: 10.1007/BF00337113. PMID 3719028